CLINICAL TRIAL: NCT06274853
Title: A Phase 1, Double-Blind, Placebo-Controlled, Randomized, Single Ascending Dose, Multiple Ascending Dose, and Food Effect Study to Assess the Safety, Tolerability, and Pharmacokinetics of GS-441524 in Healthy Subjects
Brief Title: GS-441524 for COVID-19 SAD, FE, and MAD Study in Healthy Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Operational Reasons
Sponsor: National Center for Advancing Translational Sciences (NCATS) (NIH)
Collaborators: Leidos Biomedical Research, Inc. (Industry); ICON Government and Public Health Solutions, Inc (Unknown)
Responsible Party: Sponsor
Organization: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 170327-0001; 6830/0003 (Other: ICON plc)
Record Dates: First submitted 2024-02-08; First posted 2024-02-23 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — GS-441524; stearic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- SAD Cohort 1 (Experimental): A single oral dose of 100 mg GS-441524 under fasted conditions
  Interventions: Drug: GS-441524
- SAD Placebo (Placebo Comparator): Matching Placebo under fasted conditions
  Interventions: Drug: Placebo
- SAD Cohort 2 (Experimental): A single oral dose of 300 mg GS-441524
  Interventions: Drug: GS-441524
- SAD Cohort 3 (Experimental): A single oral dose of 600 mg GS-441524
  Interventions: Drug: GS-441524
- SAD Cohort 4 (Experimental): A single oral dose of 1000 mg GS-441524
  Interventions: Drug: GS-441524
- SAD Cohort 5 (Experimental): Optional Cohort - dose TBD
  Interventions: Drug: GS-441524
- Food Effect (Experimental): Randomized, balanced, single-dose, two-treatment (fed vs fasting), two-period, two sequence crossover study part in healthy human subjects Treatment A: a single oral dose of TBD mg GS-441524 under fasted conditions Treatment B: a single oral dose of TBD mg GS-441524 under fed conditions
  Interventions: Drug: GS-441524
- MAD Cohort 1 (Experimental): Multiple oral doses of TBD mg GS-441524under fasted or fed conditions twice daily for 5 days (Days 1 to 5) and only a morning dose on Day 6
  Interventions: Drug: GS-441524
- MAD Cohort 2 (Experimental): Multiple oral doses of TBD mg GS-441524under fasted or fed conditions twice daily for 5 days (Days 1 to 5) and only a morning dose on Day 6
  Interventions: Drug: GS-441524
- MAD Cohort 3 (Experimental): Multiple oral doses of TBD mg GS-441524under fasted or fed conditions twice daily for 5 days (Days 1 to 5) and only a morning dose on Day 6
  Interventions: Drug: GS-441524
- MAD Placebo (Placebo Comparator): Matching Placebo under fasted or fed conditions
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GS-441524 — Oral GS-441524 capsules
  Other Names: (2R,3R,4S,5R)-2-(4-aminopyrrolo[2,1-f][1,2,4]triazin-7-yl)-3,4-dihydroxy-5-(hydroxymethyl)tetrahydrofuran-2-carbonitrile
  Arms: Food Effect; MAD Cohort 1; MAD Cohort 2; MAD Cohort 3; SAD Cohort 1; SAD Cohort 2; SAD Cohort 3; SAD Cohort 4; SAD Cohort 5
Drug: Placebo — Placebo capsules
  Other Names: Pregelatinized starch, colloidal silicon dioxide, magnesium stearate
  Arms: MAD Placebo; SAD Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability, and pharmacokinetics of GS-441524 in healthy subjects. The main questions to answer are: 1) What dosage of GS-441524 is required for adequate therapeutic plasma levels? 2) Does fed or fasted state produce variability in plasma levels? 3) How is GS-441524 eliminated from the body.

Participants will receive varying levels of GS-441524 or placebo to evaluate AEs and plasma levels.

DETAILED DESCRIPTION:
This study will consist of 3 parts: an a single ascending dose (SAD) part, an food effect (FE) part, and an multiple ascending dose (MAD) part.

- SAD Part This will be a randomized, double-blind, placebo-controlled single-dose study part of GS-441524 in healthy human subjects. The SAD part will consist of at least 4 cohorts and up to 5 cohorts. Subjects will be randomized into one dose cohort and receive either active drug or placebo. Within each cohort, 6 subjects will receive GS-441524 and 2 subjects will receive placebo. The proposed doses are: 100 mg, 300 mg, 600 mg, and 1000 mg.

A sentinel group of 2 subjects will be randomized to active drug or placebo (1 active; 1 placebo) and will be dosed ahead of the rest of each cohort. There will be a minimum of 48 hours between dosing of the 2 sentinel subjects and the remainder of the cohort. A review of sentinel group safety data after dosing will be completed before dose administration will continue in the remaining 6 subjects (5 active; 1 placebo) of each cohort. An optional fifth dose level may be added based on safety and PK data from the first 4 cohorts.

* FE Part This will be a randomized, balanced, single-dose, two-treatment (fed vs fasting), two-period, two sequence crossover study part in healthy human subjects using a clinically relevant dose of GS-441524 (a dose that may achieve an anticipated efficacious exposure of 2 µM3). The dose will be selected from the SAD part and will be given once under fasting conditions and once under fed conditions (after completion of a standard FDA defined high-fat breakfast) in 1 cohort of 6 subjects.
* MAD Part This will be a randomized, double-blind, placebo-controlled, repeat-dose study part of GS-441524 in healthy human subjects. There will be up to 3 dose cohorts. Subjects will be randomized into one dose cohort to receive either active drug or placebo. Within each cohort, 6 subjects will receive GS-441524 and 2 subjects will receive placebo. Subjects will be administered GS-441524 or placebo twice daily for 5 days (Days 1 to 5) and only a morning dose on Day 6.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to verbalize understanding of the consent form, able to provide written informed consent, and verbalize willingness to complete study procedures, be able to comply with protocol requirements, rules and regulations of study site, and be likely to complete all the study interventions.
* Must be considered a healthy male or healthy female of nonchildbearing potential.
* Women of nonchildbearing potential are considered women who:

  1. Do not have a uterus, or
  2. Are surgically sterile (for example: has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation; should be verified by medical documentation), or
  3. Have permanent cessation of ovarian function due to ovarian failure or surgical removal of the ovaries, or
  4. Are postmenopausal as defined by 12 months or more of spontaneous amenorrhea as confirmed by a follicle-stimulating hormone (FSH) level >30 mIU/mL.
* Between 18 and 55 years of age, inclusive.
* Body mass index (BMI) within 18.0 to 32.0 kg/m2, inclusive.
* Minimum weight of at least 50.0 kg at screening.
* Male subjects who are sexually active with female partners of childbearing potential must use, with their partner, a condom plus an approved method of effective contraception from the time of screening until 90 days after the last dose of investigational medicinal product (IMP). Additionally, male subjects must agree to not donate sperm during the study and for at least 90 days from the last dose of IMP. Effective methods of contraception are:

  1. Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal)
  2. Progestogen-only hormonal contraception (oral, injectable/implantable, or intrauterine hormone-releasing system)
  3. Implantable intrauterine device
  4. Surgical sterilization (for example, vasectomy or bilateral tubal ligation; should be verified by medical documentation)
  5. Male condom with spermicidal gel/foam or with female cap or diaphragm (double barrier)
* Must have normal renal function (estimated glomerular filtration rate [eGFR] >75 mL/min/1.73 m2, as calculated by the CKD-EPI 2021 creatinine formula).

Exclusion Criteria:

* Have a medical history of clinically significant neurological, cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, or psychiatric disorder as judged by an Investigator.
* Have clinically significant abnormal biochemistry, hematology, or urinalysis results as judged by an Investigator.
* Have disorders that may interfere with drug absorption, distribution, metabolism, and excretion processes.
* Positive test results for human immunodeficiency virus (HIV)-1/HIV-2 antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody.
* Serious cardiac illness or other medical condition including, but not limited to:

  1. Uncontrolled arrhythmias
  2. History of congestive heart failure
  3. Corrected QT value with Fridericia's formula (QTcF) >450 msec for males and >470 msec for females or history of prolonged QT syndrome
  4. Have a blood pressure reading outside of the following range: systolic blood pressure <86 mmHg or >149 mmHg and diastolic blood pressure <50 mmHg or >94 mmHg
* History of pancreatitis and history of hepatic or biliary disease, including those with known history/diagnosis of Gilbert's syndrome. Subjects with gall bladder removal <90 days prior to screening.
* Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit=12 ounces of beer, 1.5 ounces of spirit, or 5 ounces of wine) within 12 months prior to screening.
* Positive test result for alcohol and/or drugs of abuse at screening or prior to the first IMP administration.
* Current smokers and those who have smoked within 90 days prior to the first IMP administration. Current users of e cigarettes and nicotine replacement products, and those who have used these products within 90 days prior to the first IMP administration.
* Concurrent treatment or treatment with an investigational drug within 30 days prior to the first dose of IMP.
* Blood donation of approximately 500 mL within 56 days or plasma donation within 7 days of screening.
* Subjects who are taking, or have taken, any prescribed or over-the-counter drugs (other than a maximum of 2 g per day of acetaminophen, hormone replacement therapy, hormonal contraception) or herbal remedies in the 14 days before randomization. Exceptions may apply on a case-by-case basis if considered not to interfere with the objectives of the study, as agreed by the Investigator and Sponsor's Medical Monitor.
* Known allergy or intolerance to remdesivir.
* Any condition that, in the opinion of an Investigator, would interfere with evaluation or interpretation of subject safety or study results.
* Affiliated with, or a family member of, site staff directly involved in the study, or anyone with a financial interest in the outcome of the study.
* Subjects who are unable, in the opinion of an Investigator, to comply fully with the study requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) | 10 days
  Number of incidences
Blood Pressure in mm/Hg | 10 days
  Changes from baseline
Pulse in beats/min | 10 days
  Changes from baseline
Respiratory Rate in breaths per minute | 10 days
  Changes from baseline
Body Temperature in degrees | 10 days
  Changes from baseline
Electrocardiogram (ECG) as measured by PR interval | 10 days
  Changes from baseline
Electrocardiogram (ECG) as measured by QT interval | 10 days
  Changes from baseline
Electrocardiogram (ECG) as measured by QT corrected (Fridericia's) | 10 days
  Changes from baseline

SECONDARY OUTCOMES:
Plasma PK Parameter C-Max | 10 days
  Maximum observed plasma concentration
Plasma PK Parameter t-max | 10 days
  Time to attain maximum observed plasma concentration
Plasma PK Parameter t-lag | 10 days
  Time before the first concentration above the lower limit of quantitation
Plasma PK Parameter AUC 0-last | 6 days
  Area under the plasma concentration time curve from time zero to the last quantifiable time point
Plasma PK Parameter AUC 0-inf | 6 days
  Area under the plasma concentration time curve from time 0 to infinity
Plasma PK Parameter t 1/2 | 10 days
  Terminal elimination half-life
Plasma PK Parameter CL/F | 10 days
  Apparent oral clearance
Plasma PK Parameter Vz/F | 10 days
  Apparent volume of distribution
Urine PK Parameter Ae urine | 10 days
  Cumulative amount of study drug excreted in urine
Urine PK Parameter Fe urine | 10 days
  Fraction of the dose administered excreted (unchanged in urine)
Urine PK Parameter CL R | 10 days
  Renal clearance
Plasma PK Parameter C trough | 10 days
  Trough Plasma concentration
Plasma PK Parameter AUC 0-tau | 10 days
  Area under the plasma concentration time curve over a dosing interval tau
Plasma PK Parameter CL/F ss | 10 days
  Apparent oral clearance at steady state
Plasma PK Parameter Vz/F ss | 10 days
  Apparent volume of distribution at steady state
Plasma PK Parameter R ac | 10 days
  Accumulation ration, based on Auc 0-tau of day 6 versus day1

CONTACTS AND LOCATIONS:
Overall Officials: Philip E Sanderson, PhD, Study Director — NCATS

IPD SHARING:
Plan to Share IPD: No